CLINICAL TRIAL: NCT05361096
Title: The Effect of Flipped Learning Approach on Nursing Students' Learning of Patient Safety: A Mixed Methods Study
Brief Title: The Effect of Flipped Learning Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, Principal investigator (Dr. Research Assistant), Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GaziU-SBF-EE-01
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: nursing education

STUDY DESIGN:
Intervention Model Description: Explanatory sequential design, one of the mixed-method designs, was used.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational approach (Flipped learning) group (Experimental): The teaching of the patient safety subject was performed with the flipped learning to the intervention group (n=45).
  Interventions: Other: Educational approach (Flipped learning)
- Traditional education group (No Intervention): The teaching of the patient safety subject was performed with the traditional educational to the control group (n=44).

INTERVENTIONS:
Other: Educational approach (Flipped learning) — In the intervention group, the out-of-class stage started one week before the in-class stage of the relevant week. The researchers covered the topic of the week asynchronously in the virtual classroom in the learning management system. Students have been able to log into the system at anytime and anywhere and study the course video and other course materials repeatedly.
  The in-class stage is the session in which the students in the intervention group come together with the researcher synchronously and conduct an online lesson. It was conducted one session per week for four weeks. The course was carried out synchronously on the Zoom platform during the in-class stage.
  Arms: Educational approach (Flipped learning) group

SUMMARY:
This study was conducted to evaluate the effect of flipped learning approach on nursing students' learning of patient safety.

DETAILED DESCRIPTION:
Patient safety is the basis of all theoretical and practical subjects in nursing. In the literature, while the traditional approach in nursing education has been stated to be insufficient in developing knowledge, attitudes and skills related to patient safety , the flipped learning approach is considered to be effective. During the out-of-class stage of the flipped learning approach, using the practices such as showing videos related patient safety, enriching course presentations and videos with interactive questions, organizing discussion sessions on forum pages and sharing educational games contribute to the students' following the subject more carefully. In the in-class stage, the use of activities such as case studies, group discussions, simulation, concept maps, various interactive methods and active participation of students in these activities is important. Teaching methods appealing to different learning styles and senses make it easier to look at the subject from different perspectives and establish a cause-effect relationship.

The evaluation of learning outcomes related to patient safety with the flipped learning approach is thought to provide guidance to nursing students and educators in terms of learning and teaching experiences.

The teaching of the patient safety subject was performed with the traditional educational to the control group (n=44) and with the flipped learning to the intervention group (n=45). Quantitative and quantitative data were collected with the "Demographic information form", "Achievement test", "Patient safety competency self-evaluation scale", and "Semi-structured focus group interview form". Quantitative data were collected before the applications, when the applications were completed, and six weeks after the applications. When the flipped learning approach was completed, qualitative data were collected.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in the Nursing Fundamentals II Course for the first time,
* Sufficient or unlimited internet access,
* Accepting to process the simultaneous lessons of patient safety on the Zoom platform,
* Being willing to participate in the research.

Exclusion Criteria:

* Having a high school, associate or undergraduate degree in a health-related field,
* To have taken a course on patient safety before.
* The student's desire to leave the research at any stage,
* Not filling in data collection forms.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Development of cognitive knowledge about patient safety | After the completion of the 4-week patient safety course, the achievement test (post-test) was administered to both groups immediately. After 6 weeks, the change in the knowledge level of the groups was measured again with the test (follow-up).
  The achievement test prepared by the researchers according to the literature. It consists of 20 questions each with five options to measure the knowledge level for patient safety. These questions were on general knowledge (4 questions), identify patients correctly (2 questions), safe drug administration (6 questions), fall (5 questions), and infection (3 questions). An increase in the score from the test indicates a high level of knowledge about patient safety (min: 0 point, max: 100 point).
Development of patient safety competency | Patient Safety Competency Self-Evaluation Scale was applied immediately for both of the groups after the course, which lasted for 4 weeks, was completed. After 6 weeks, the change in the self-assesment of the groups was measured again with the scale.
  Patient Safety Competency Self-Evaluation Scale is a valid and reliable data collection scale. The scale, a five-point Likert type, has 36 items. It consists of three categories: knowledge, skills, and attitude. An increase in the score from the scale indicates an increase in competencies related to patient safety. (With a minimum potential score of 36 and a maximum score of 180). The Cronbach alpha coefficient was 0.95.
Determining students' views on patient safety | Immediately after flipped learning approach was completed, qualitative data were collected.
  The semi-structured focus group interview form was developed by the researchers. The researchers designed these questions on the basis of both their experiences and the literature. It consists of six open-ended questions in which students share their opinions on the flipped learning approach. Focus group discussions were conducted of students in the intervention group. A total of 25 students who volunteered to participate in the interviews were selected.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Eyikara, Principal Investigator — Doctor Research assistant
Locations (1):
- Gazi University Department of Health Sciences, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No